CLINICAL TRIAL: NCT06823440
Title: Prevention of Chemotherapy-induced Polyneuropathy (CIPN) Using Compressive Therapy
Brief Title: Prevention of CIPN Using Compressive Therapy
Acronym: CIPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martina Lojova (Other)
Responsible Party: Sponsor-Investigator, Martina Lojova, Tatiana Ciprova, lead nurse, Department of Comprehensive Cancer Care, Masaryk Memorial Cancer Institute, Brno, Czech Republic., Masaryk Memorial Cancer Institute
Organization: Masaryk Memorial Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOU-2024-03
Record Dates: First submitted 2025-01-31; First posted 2025-02-12 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: CIPN in Adjuvant Breast Cancer Patients
Keywords: CIPN; breast cancer; compressive therapy; chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A - compression short (Experimental): In Arm A, patients will wear compression gloves beginning 15 min before the start of paclitaxel infusion, during infusion, and for 30 min post-paclitaxel infusion. They will also wear the compression knee socks beginning 15 minutes before the start of paclitaxel infusion, during infusion, and for 90 minutes post-paclitaxel infusion.
  Interventions: Device: Compression using surgical gloves and compression knee socks
- B - compression long (Experimental): In Arm B, patients will wear compression gloves beginning 15 min before the start of paclitaxel infusion, during infusion, and for 90 minutes post-paclitaxel infusion. They will also wear the compression knee socks beginning 15 minutes before the start of paclitaxel infusion, during infusion, and for 24 hours post-paclitaxel infusion.
  Interventions: Device: Compression using surgical gloves and compression knee socks
- C - no compression (No Intervention): Nonrandomized control group with no compression intervention.

INTERVENTIONS:
Device: Compression using surgical gloves and compression knee socks — Compression therapy will be applied using surgical gloves and compression knee socks. The compression itself will take place on the principle of compressing the limbs, which will narrow the blood vessels and thereby limit the flow of cytostatics to the peripheral parts of the body. This is believed to reduce damage to nerve fibers. Special knee socks with compression of 20-30 mm Hg and latex/nitrile surgical gloves will be used for pressure therapy. The size of the compression aids will be determined by the nursing staff (gloves will be a tight-fitting size; they will not cause discomfort). The patients will wear the compression aids for a specific amount of time before administering paclitaxel, throughout paclitaxel infusion, and after the infusion.
  Arms: A - compression short; B - compression long

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common side effect of treatment with taxanes and platinum-based drugs, significantly impacting the quality of life of oncology patients. Symptoms such as reduced sensitivity and pain may persist even after treatment ends. Research has shown that compression therapy using gloves and stockings effectively reduces the incidence of CIPN, improves patient adherence to treatment, and has no severe side effects. A study at the Chemotherapy Unit of the Comprehensive Oncology Care Clinic, Masaryk Memorial Cancer Institute, will investigate the efficacy of this therapy. Tight-fitting gloves and compression stockings will be used to limit the flow of cytotoxic agents to peripheral areas. Effectiveness will be assessed through quality-of-life questionnaires, hand strength and coordination tests, and laboratory analyses to identify predictive markers of neuropathy. The study aims to enhance CIPN prevention and integrate this method into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years at the time of signing the informed consent (IC).
* Signed informed consent.
* Breast cancer stages I-III
* ECOG performance status 0-2.
* (Neo)adjuvant treatment with paclitaxel weekly.

Exclusion Criteria:

* Metastatic disease.
* History of neuropathy/vasculopathy and its pharmacological treatment.
* Type I or II diabetes.
* Stroke within the last 6 months.
* Prior treatment with taxanes and/or cisplatin derivatives.
* Peripheral arterial ischemia.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in reported EORTC QLQ CIPN20 subscales | Before paclitaxel course (baseline) and completion paclitaxel course (standardly 12 weeks)
  The preventive effect of compression therapy will be evaluated based on changes reported in a survey, using self-reported neuropathy assessed with EORTC QLQ-CIPN 20, which contains 20 items divided into three subscales assessing sensory, motor, and autonomic symptoms. Each item is scored on a Likert scale ranging from 1 (not at all) to 4 (very much). Scores will be converted to a 0-100 scale, with higher scores representing more higher scores represent more symptoms/problems.

SECONDARY OUTCOMES:
Changes in reported EORTC QLQ-C30 subscales | Before paclitaxel course (baseline), after the sixth cycle of paclitaxel (standardly 6 weeks), after completion paclitaxel course (standardly 12 weeks) and six months after completition paclitaxel course
  QoL will be assessed with the EORTC QLQ-C30, which contains 30 items. Each item is scored on a Likert scale ranging from 1 (not at all) to 4 (very much), except for the global QoL scale that ranges from 1 (very poor) to 7 (excellent). The item will be transformed into a global health status (GHS) scale, five functional scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, pain, and nausea-vomiting), and six single-item symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Scores will be converted to a 0-100 scale. Higher numerical scores on functional scales or the GHS scale indicate better QoL, while higher scores on symptom scales/items reflect a greater level of symptoms or problems.
Changes in reported EORTC QLQ CIPN20 subscales | Before paclitaxel course (baseline), after the sixth cycle of paclitaxel (standardly 6 weeks), after completion paclitaxel course (standardly 12 weeks) and six months after completition paclitaxel course
  The preventive effect of compression therapy will be evaluated based on changes reported in a survey, using self-reported neuropathy assessed with EORTC QLQ-CIPN 20, which contains 20 items divided into three subscales assessing sensory, motor, and autonomic symptoms. Each item is scored on a Likert scale ranging from 1 (not at all) to 4 (very much). Scores will be converted to a 0-100 scale, with higher scores representing more higher scores represent more symptoms/problems.

OTHER OUTCOMES:
Changes in hand grip test a grip ability test | Before paclitaxel course (baseline), after the sixth cycle of paclitaxel (standardly 6 weeks), after completion paclitaxel course (standardly 12 weeks) and six months after completition paclitaxel course
  In the Hand grip test, the hand grip strength is measured three times for each upper limb with a rest interval between each grip of the device handle. The grip ability test is a modification of the general hand function test based on daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Ciprova, MBA, Principal Investigator — Masaryk Memorial Cancer Institute
Locations (1):
- Masaryk Memorial Cancer Institute, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No